CLINICAL TRIAL: NCT06488703
Title: Retrospective Analysis of Systemic Glucocorticoid Mediated Long-term Effects, Patient Pathways and Economic Burden Across Multiple Indications [PROGRESS Study]
Brief Title: Retrospective Analysis of Systemic Glucocorticoid Mediated Long-term Effects, Patient Pathways and Economic Burden Across Multiple Indications
Status: Active, not recruiting | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Vandage GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 222292
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: PROGRESS; Systemic (cortico)steroids / systemic glucocorticoids; Long term OCS side effects; OCS side effects; SCS side effects; Long term SCS side effects; Asthma; Chronic obstructive pulmonary disease (COPD); Rheumatism; Lupus; Vasculitis; Eosinophilic granulomatosis with polyangiitis (EGPA); Chronic rhinosinusitis with nasal polyps (CRSwNP); Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Rheumatic Diseases; Vasculitis; Churg-Strauss Syndrome; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Participants with underlying condition (UC): Participants with UCs (Bronchial Asthma, coronary obstructive pulmonary disorder [COPD], Chronic Arthritis und Rheumatism, Systemic lupus erythematosus, Vasculitis, Eosinophilic granulomatosis with polyangiitis [EGPA], Chronic rhinosinusitis [CRS], Crohn's disease, and Ulcerative colitis) with Systemic (cortico)steroids/systemic glucocorticoids (SCS) exposure will be evaluated.
- Matching control group: Participants with the same UC but without SCS treatment will be evaluated.

SUMMARY:
Glucocorticoids are important in the treatment of many inflammatory, allergic, immunologic, and malignant disorders. However, the adverse effects of systemic corticosteroids are one of the most common causes of iatrogenic conditions associated with chronic inflammatory diseases. Limited data are available about long-term- Systemic (cortico)steroids / systemic glucocorticoids (SCS) related side effects. Oral (cortico)steroids / systemic glucocorticoids (OCS) mediated side effects in e.g., rheumatic diseases are not consistently determined. No sufficient cohort analysis determined systematically possible side effects of SCS in the long-term. This study will close this major gap by delivering data about long-term SCS side effects (risk stratification via SCS dose, treatment duration). Therefore, the primary objective of PROGRESS is to quantify the risk of adverse outcomes among populations with specific underlying conditions (UC) with and without exposition to systemic glucocorticoid therapy in Germany. The secondary objective is to analyze the influence of dosage and time of systemic glucocorticoid therapy exposition on the risk of adverse outcomes among these populations with specific UCs. In general, it is evident that a frequent SCS exposure leads to side effects like diabetes or osteoporosis etc., which have the potential to become a major financial burden to healthcare systems. For this reason, the tertiary objective is to quantify the economic burden associated with the incidence of adverse outcomes related to SCS exposition among populations with specific UCs for the German market. The study design will be a retrospective cohort study (claims data) based on a rolling cohort design using an exact matching approach. Persons with different UCs and with SCS treatment exposition are matched to controls with UC but without SCS treatment. Matching will be performed on a quarterly basis. First patient-in is in 01/2009, last patient-in in 12/2020. The study period covers data from 01/2007 to 12/2022. The study population are adult patients with confirmed diagnosis of Bronchial Asthma, COPD, Chronic Arthritis und Rheumatism, Systemic lupus erythematosus, Vasculitis, Eosinophilic granulomatosis with polyangiitis (EGPA), Chronic rhinosinusitis (CRS), Crohn's disease, or Ulcerative colitis in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older.
* Prevalent diagnosis of an underlying condition.
* At least two years of pre observation period. The same inclusion criteria apply to the matched control group, excluding the initiation of Systemic (cortico)steroids / systemic glucocorticoids (SCS) treatment.

Exclusion Criteria:

* Have a record of defined SCS-related adverse outcome within two years before index date.
* Have a history of breast cancer and / or tamoxifen prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll participants who meets the below inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 52000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with specific Adverse outcome in patients with underlying condition (UC) with exposition of systemic glucocorticoids | Up to 7 months
  Percentage of participants with specific adverse outcome among participants with UC with exposition of systemic glucocorticoids will be assessed. Specific adverse outcomes includes incident diagnosis of Type 2 diabetes mellitus, Malignant neoplasm of bladder, non-Hodgkin lymphoma, Cardio-/cerebrovascular disease, Myocardial infarction, Atrial fibrillation and flutter, Heart failure, Cerebrovascular accident, Dyslipidemia, Hypertension, Obesity / abnormal weight gain, Osteoporosis, Osteoporosis diagnosis with osteoporotic fractures, Glaucoma, Cataract, Peptic ulcer, Acute mental disorder, Sleep disorders, Pneumonia, Musculoskeletal disorders, Sepsis, Cystitis, Gastric ulcer, or Functional dyspepsia.
Percentage of Participants with any Adverse outcome in patients with underlying condition (UC) with exposition of systemic glucocorticoids | Up to 7 months
  Percentage of participants with any adverse outcome among participants with UC with exposition of systemic glucocorticoids will be assessed. Specific adverse outcomes includes incident diagnosis of Type 2 diabetes mellitus, Malignant neoplasm of bladder, non-Hodgkin lymphoma, Cardio-/cerebrovascular disease, Myocardial infarction, Atrial fibrillation and flutter, Heart failure, Cerebrovascular accident, Dyslipidemia, Hypertension, Obesity / abnormal weight gain, Osteoporosis, Osteoporosis diagnosis with osteoporotic fractures, Glaucoma, Cataract, Peptic ulcer, Acute mental disorder, Sleep disorders, Pneumonia, Musculoskeletal disorders, Sepsis, Cystitis, Gastric ulcer, or Functional dyspepsia.
Percentage of Participants with specific Adverse outcome in participants with UC without exposition of systemic glucocorticoids | Up to 7 months
  Percentage of participants with specific adverse outcome among participants with UC without exposition of systemic glucocorticoids will be assessed. Specific adverse outcomes includes incident diagnosis of Type 2 diabetes mellitus, Malignant neoplasm of bladder, non-Hodgkin lymphoma, Cardio-/cerebrovascular disease, Myocardial infarction, Atrial fibrillation and flutter, Heart failure, Cerebrovascular accident, Dyslipidemia, Hypertension, Obesity / abnormal weight gain, Osteoporosis, Osteoporosis diagnosis with osteoporotic fractures, Glaucoma, Cataract, Peptic ulcer, Acute mental disorder, Sleep disorders, Pneumonia, Musculoskeletal disorders, Sepsis, Cystitis, Gastric ulcer, or Functional dyspepsia.
Percentage of Participants with any Adverse outcome in participants with UC without exposition of systemic glucocorticoids | Up to 7 months
  Percentage of participants with any adverse outcome among participants with UC without exposition of systemic glucocorticoids will be assessed. Specific adverse outcomes includes incident diagnosis of Type 2 diabetes mellitus, Malignant neoplasm of bladder, non-Hodgkin lymphoma, Cardio-/cerebrovascular disease, Myocardial infarction, Atrial fibrillation and flutter, Heart failure, Cerebrovascular accident, Dyslipidemia, Hypertension, Obesity / abnormal weight gain, Osteoporosis, Osteoporosis diagnosis with osteoporotic fractures, Glaucoma, Cataract, Peptic ulcer, Acute mental disorder, Sleep disorders, Pneumonia, Musculoskeletal disorders, Sepsis, Cystitis, Gastric ulcer, or Functional dyspepsia.

SECONDARY OUTCOMES:
Percentage of Participants with specific Adverse outcome in the influence of systemic glucocorticoid therapy exposition related to dosage and time. | Up to 7 months
  Percentage of participants with specific adverse outcome in the influence of systemic glucocorticoid therapy exposition related to dosage and time will be assessed. Specific adverse outcomes includes incident diagnosis of Type 2 diabetes mellitus, Malignant neoplasm of bladder, non-Hodgkin lymphoma, Cardio-/cerebrovascular disease, Myocardial infarction, Atrial fibrillation and flutter, Heart failure, Cerebrovascular accident, Dyslipidemia, Hypertension, Obesity / abnormal weight gain, Osteoporosis, Osteoporosis diagnosis with osteoporotic fractures, Glaucoma, Cataract, Peptic ulcer, Acute mental disorder, Sleep disorders, Pneumonia, Musculoskeletal disorders, Sepsis, Cystitis, Gastric ulcer, or Functional dyspepsia.
Percentage of Participants with any Adverse outcome in the influence of systemic glucocorticoid therapy exposition related to dosage and time. | Up to 7 months
  Percentage of participants with any adverse outcome in the influence of systemic glucocorticoid therapy exposition related to dosage and time will be assessed.
Percentage of Participants with any Adverse outcome in the influence of systemic glucocorticoid therapy without exposition related to dosage and time. | Up to 7 months
  Percentage of participants with any adverse outcome in the influence of systemic glucocorticoid therapy exposition related to dosage and time will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Rwth Aachen University-Aachen-Germany-C, Germany, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/